CLINICAL TRIAL: NCT00621036
Title: A Phase 2, Open-Label Study to Evaluate the Efficacy and Safety of Patient-Specific Immunotherapy, Recombinant Idiotype Conjugated to KLH (Id-KLH) and Administered With GM-CSF, in Patients With CNS Lymphoma
Brief Title: Vaccine Therapy and GM-CSF in Treating Patients With CNS Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: MyVax did not meet its primary endpoints
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-02F07; SCCC-102007-035; CDR0000587504 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-02-21; First posted 2008-02-22 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma; Lymphoproliferative Disorder; Small Intestine Cancer
Keywords: primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; stage IV adult T-cell leukemia/lymphoma; adult nasal type extranodal NK/T-cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; intraocular lymphoma; post-transplant lymphoproliferative disorder; cutaneous B-cell non-Hodgkin lymphoma; Waldenström macroglobulinemia; small intestine lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Lymphoproliferative Disorders; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Intraocular Lymphoma; Waldenstrom Macroglobulinemia | interventions — sargramostim; Methotrexate; Thiotepa; Radiotherapy

ARMS (1):
- methotrexate IV once every 2 weeks (Experimental)
  Interventions: Biological: autologous immunoglobulin idiotype-KLH conjugate vaccine; Biological: sargramostim; Drug: methotrexate; Drug: thiotepa; Radiation: radiation therapy

INTERVENTIONS:
Biological: autologous immunoglobulin idiotype-KLH conjugate vaccine
Biological: sargramostim
Drug: methotrexate
Drug: thiotepa
Radiation: radiation therapy

SUMMARY:
RATIONALE: Vaccines made from a person's cancer proteins may help the body build an effective immune response to kill cancer cells. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving vaccine therapy together with GM-CSF may make a stronger immune response and kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects and how well giving vaccine therapy together with GM-CSF works in treating patients with CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the proportion of patients with CNS lymphoma who develop anti-idiotype (Id) and anti-keyhole limpet hemocyanin (KLH) humoral immune responses in the serum and/or CSF following patient-specific immunotherapy comprising recombinant tumor-derived immunoglobulin Id-KLH conjugate vaccine and sargramostim (GM-CSF).
* To assess the safety and tolerability of this regimen in these patients.

Secondary

* To evaluate the progression-free survival (PFS) of patients treated with this regimen.
* To determine the time to receipt of first subsequent anti-lymphoma therapy after initiating immunization with the Id-KLH conjugate vaccine.
* To assess the correlation of anti-Id immune response in the CSF and/or serum with PFS and overall survival.

Tertiary

* To evaluate the kinetics of humoral immune response development in patients treated with this regimen.

OUTLINE:

* Pre-immunotherapy: Patients submit a tumor sample for manufacturing of the idiotype (Id)-keyhole limpet hemocyanin (KLH) conjugate vaccine and undergo placement of an Ommaya reservoir. Patients then receive induction therapy comprising methotrexate IV once every 2 weeks until a maximum radiographic response is achieved, as assessed by MRI of the brain. Patients then receive methotrexate IV once a month for 6 months. Patients with leptomeningeal or CSF involvement also receive intraventricular thiotepa twice a week until the CSF is clear on three evaluations and then once a week until the CSF is clear on four evaluations. Patients under 55 years of age also undergo whole brain radiotherapy (or craniospinal radiotherapy when extensive leptomeningeal disease is present). Patients who achieve a stable response to induction therapy proceed to immunotherapy.
* Immunotherapy: Patients receive recombinant tumor-derived immunoglobulin Id-KLH conjugate vaccine subcutaneously (SC) on day 1 of weeks 0, 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, and 76. Patients also receive sargramostim (GM-CSF) SC on days 1-4 of the same weeks as the Id-KLH conjugate vaccine.

After completion of therapy, patients are followed periodically for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or CSF cytologically confirmed CNS lymphoma with any of the following clinical histories:

  * Primary CNS lymphoma at initial diagnosis
  * Primary CNS lymphoma at relapse
  * Systemic lymphoma with CNS disease at initial diagnosis or at relapse
* Adequate fresh tissue or cell pellet available for analysis by Genitope Corporation to determine adequacy for idiotype (Id) manufacturing
* Tumor must express both functional light and heavy chain genes
* No tumors known or found to be surface immunoglobulin negative
* Not in leukemic phase (i.e., > 5,000/mm³ circulating tumor cells)

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 70-100%
* WBC ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin ≥ 10 g/dL
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN) (unless due to Gilbert's disease)
* Creatinine ≤ 1.5 times ULN
* Able to undergo placement of an Ommaya reservoir
* Able to receive induction therapy (chemotherapy with or without brain radiotherapy) with intent to induce remission
* Speaks English or Spanish
* No other malignancy within the past 3 years, except adequately treated basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ
* Not pregnant or nursing
* No immunosuppressive viral infections as evidenced by HIV antibody or antigen, hepatitis B antigen, or hepatitis C antibody or antigen positivity
* No history of autoimmune disease that required treatment within the past 5 years, including previously treated autoimmune hemolytic anemia or immune thrombocytopenia

PRIOR CONCURRENT THERAPY:

* More than 30 days since prior and no concurrent participation in another therapeutic clinical trial
* More than 2 weeks since prior steroids
* No concurrent immunosuppressives, including corticosteroids

  * Transient use of optical or nasal steroid solutions is allowed
* No other concurrent anticancer therapy or therapy for non-Hodgkin lymphoma

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10-19 (Actual); Primary Completion 2008-12-08 (Actual); Study Completion 2008-12-08 (Actual)

PRIMARY OUTCOMES:
Anti-idiotype (Id) and anti-keyhole limpet hemocyanin (KLH) immune response rate in the CSF
Safety and tolerability

SECONDARY OUTCOMES:
Progression-free survival (PFS)
Time to receipt of first subsequent anti-lymphoma therapy after initiating immunization with the Id-KLH conjugate vaccine
Correlation of anti-Id immune response in the CSF and/or serum with PFS and overall survival
Kinetics of humoral immune response development

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Maher, MD, PhD, Principal Investigator — Simmons Cancer Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States